CLINICAL TRIAL: NCT06710106
Title: Effect of a Low-calorie Diet With a Prebiotic Supplement on Health of Overweight-obese Subjects: a Randomized Controlled Trial
Brief Title: Effect of a Low-calorie Diet With a Prebiotic Supplement on Health of Overweight-obese Subjects.
Acronym: POSTBIOTICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POSTBIOTICS (2024.154)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Polyphenols; Obesity; Weight Loss
Keywords: supplement; obesity; polyphenols; prebiotic; microbiota
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Parallel groups, blind, 8-week randomized nutritional intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prebiotic group (Experimental): Natural yogurt with prebiotic formula
  Interventions: Dietary Supplement: Prebiotic + hypocaloric diet
- Placebo group (Placebo Comparator): Natural yogurt with placebo formula
  Interventions: Dietary Supplement: Placebo + hypocaloric diet

INTERVENTIONS:
Dietary Supplement: Prebiotic + hypocaloric diet — Study participants will add prebiotic formula in a natural yogurt every day to be consumed within a hypocaloric diet.
  Arms: Prebiotic group
Dietary Supplement: Placebo + hypocaloric diet — Study participants will add placebo formula in a natural yogurt every day to be consumed within a hypocaloric diet.
  Arms: Placebo group

SUMMARY:
The main objective of this project is to evaluate the effect of prebiotic supplementation on weight loss and other physiological and metabolic parameters related to excess weight in overweight/obese adult men and women, as well as to determine the changes in the gut microbiota associated with these changes. Specific objectives are focus on evaluate the effect of the intervention on the following parameters:

* Weight and body composition.
* Changes in the gut microbiota (metagenomics).
* Changes in urinary and serum metabolites.
* Complete blood count, routine biochemical variables related to glucose and lipid metabolism, as well as liver health parameters.
* Specific markers involved in obesity pathology (insulin, leptin, adiponectin, and cytokines MCP1, TNF, CRP, and IL10).
* Satiety-related variables using a visual analog scale.
* Adherence to the assigned intervention, both to the hypocaloric diet and to the supplement provided in the study.
* Physical activity level.
* Changes in gastrointestinal health through self-reported questionnaires.
* Mental health and quality of life of participants through self-reported questionnaires.
* Chronotype of participants through a self-reported questionnaire. For this purpose, a randomized, double blind parallel study has been designed.

Target sample size is 156 subjects.

Participants will be allocated in two groups for 8 weeks:

* Experimental group (n=104): hypocaloric diet + prebiotic supplement.
* Placebo group (n=52): hypocaloric diet + placebo supplement.

Participants will visit nutritional intervention unit at week 1 and week 8. At week 4 they will receive a phone control call.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will be interviewed by phone to verify that they meet the main inclusion criteria. Volunteers who meet the main inclusion criteria will be invited to an information and screening visit to resolve any doubts. Volunteers who agree to participate in the study will sign the informed consent and will be randomly allocated to one of the two arms of the study and will be provided with any required material.

During the intervention, volunteers will attend 2 Clinical investigation visits. The first one will be carried out on the first day of the study and the last one will take place at the end of the 8 weeks. In both visits anthropometric and body composition measurements, blood pressure, stool and blood, urine and stool samples, as well as data about dietary, physical activity, sleep and gastrointestinal symptoms will be taken.

Inclusion criteria

* Men and women aged 18 to 70 years.
* Volunteers with overweight or obesity (BMI: 25.0-39.9 kg/m²) and body fat percentage > 30% for women / > 20% for men.
* Stable weight (+/- 5%) in the last three months prior to the start of the study.
* Normal physical examination and vital signs, or clinically insignificant findings for the experiment (those not related to metabolic health).
* Subjects must be able to understand and be willing to sign the informed consent form, agreeing to comply with all study procedures and requirements.
* Continued pharmacological/hormonal treatment will be allowed as long as it does not affect the study parameters and the dosage has been stable for at least 3 months. Exclusion will apply to treatments with insulin or any drug with hypoglycemic effects.
* Willingness to undergo each of the procedures involved in the study (including consuming a sweetened yogurt).
* Availability to attend the two in-person clinical evaluation sessions at the scheduled times and locations.

Exclusion criteria

* Volunteers undergoing pharmacological treatment if the treatment is not stable (at least 3 months before the start of the study), with exclusion of treatments:
* That alter gastrointestinal function.
* Stomach protectants.
* Hypoglycemic drugs.
* Insulin (under no circumstances).
* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects who have undergone surgical interventions with permanent sequelae in the digestive system (e.g., gastroduodenostomy) or bariatric surgery.
* Suffering from any chronic metabolic disease or obesity-related disease, or any systemic intestinal, liver, or kidney disease: type 1 or 2 diabetes, severe dyslipidemia, uncontrolled thyroid dysfunction, cirrhosis, inflammatory bowel disease, untreated anemia, etc. (non-alcoholic fatty liver will not be an exclusion criterion).
* Exceeding the alcohol consumption limit for the corresponding sex (more than 14 units per week for women and 20 units per week for men).
* Pregnant, breastfeeding, or planning to become pregnant.
* Taking nutritional supplementation (weight loss supplements, fiber supplements, probiotics, multivitamins, etc.) that contains compounds that may affect the study outcomes, unless the person is willing to stop these supplements during the 8-week intervention period and ensures a minimum washout period of 30 days before baseline measurements.
* Having donated blood in the 14 days prior to the start visit.
* Subjects with any type of cancer or undergoing cancer treatment, or who have not been free of cancer for at least 5 years since eradication.
* Subjects with an allergy to any component of the study product or any other food that interferes with and complicates following the study protocol.
* Subjects with any cognitive and/or psychiatric impairment.
* Subjects who are expected to have poor cooperation or, in the investigator's opinion, have difficulty following the study procedures.
* Subjects currently undergoing treatment for weight loss/body composition modification.
* Subjects who are taking or have taken antibiotics within 30 days before the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 70 years.
* Volunteers with overweight or obesity (BMI: 25.0-39.9 kg/m²) and body fat percentage > 30% for women / > 20% for men.
* Stable weight (+/- 5%) in the last three months prior to the start of the study.
* Normal physical examination and vital signs, or clinically insignificant findings for the experiment (those not related to metabolic health).
* Subjects must be able to understand and be willing to sign the informed consent form, agreeing to comply with all study procedures and requirements.
* Continued pharmacological/hormonal treatment will be allowed as long as it does not affect the study parameters and the dosage has been stable for at least 3 months. Exclusion will apply to treatments with insulin or any drug with hypoglycemic effects.
* Willingness to undergo each of the procedures involved in the study (including consuming a sweetened yogurt).
* Availability to attend the two in-person clinical evaluation sessions at the scheduled times and locations.

Exclusion Criteria:

* Volunteers undergoing pharmacological treatment if the treatment is not stable (at least 3 months before the start of the study), with exclusion of treatments:
* That alter gastrointestinal function.
* Stomach protectants.
* Hypoglycemic drugs.
* Insulin (under no circumstances).
* Subjects with relevant functional or structural abnormalities of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux, etc.
* Subjects who have undergone surgical interventions with permanent sequelae in the digestive system (e.g., gastroduodenostomy) or bariatric surgery.
* Suffering from any chronic metabolic disease or obesity-related disease, or any systemic intestinal, liver, or kidney disease: type 1 or 2 diabetes, severe dyslipidemia, uncontrolled thyroid dysfunction, cirrhosis, inflammatory bowel disease, untreated anemia, etc. (non-alcoholic fatty liver will not be an exclusion criterion).
* Exceeding the alcohol consumption limit for the corresponding sex (more than 14 units per week for women and 20 units per week for men).
* Pregnant, breastfeeding, or planning to become pregnant.
* Taking nutritional supplementation (weight loss supplements, fiber supplements, probiotics, multivitamins, etc.) that contains compounds that may affect the study outcomes, unless the person is willing to stop these supplements during the 8-week intervention period and ensures a minimum washout period of 30 days before baseline measurements.
* Having donated blood in the 14 days prior to the start visit.
* Subjects with any type of cancer or undergoing cancer treatment, or who have not been free of cancer for at least 5 years since eradication.
* Subjects with an allergy to any component of the study product or any other food that interferes with and complicates following the study protocol.
* Subjects with any cognitive and/or psychiatric impairment.
* Subjects who are expected to have poor cooperation or, in the investigator's opinion, have difficulty following the study procedures.
* Subjects currently undergoing treatment for weight loss/body composition modification.
* Subjects who are taking or have taken antibiotics within 30 days before the initial visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fecal microbiota of participants will be analyzed by bacterial 16S or Shotgun gene sequencing technology.

SECONDARY OUTCOMES:
Body weight | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body mass index will be calculated as follows: weight (kilograms)/ height (cm)2
Body fat percentage | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body fat of participants will be analyzed by bioimpedance and reported in percentage and kilograms.
Body muscle mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body muscle mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body lean mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body leen mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body water mass | Clinical Investigation Day 1 and Clinical Investigation Day 2.]
  Body water mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body bone mass | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Body bone mass of participants will be analyzed by bioimpedance and reported in kilograms.
Gastrointestinal symptoms | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Gastrointestinal symptoms will be registrated through Gastrointestinal Symptoms Rating Scale questionnaire, which is a questionnaire of 15 items. The questionnaire has a seven-point graded likert-type scale, where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Dietary intake | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Dietary intake (energy, macronutrients and micronutrients) will be analysed by food frequency questionnaire.
Physical activity | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Physical activity will be evaluated by the reduced version of the International Physical Activity Questionnaire, which estimates the total physical activity in MET-min/week, time spent sitting and classifies subjects based on their physical activity
Adherence to capsule consumption | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Adherence will be assessed using the capsule consumption record form.
Waist circumference | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Waist circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Hip circumference | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Hip circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Neck circumference | linical Investigation Day 1 and Clinical Investigation Day 2
  Neck circumference of participants in fasting condition will be analyzed by measuring tape and reported in centimeters.
Systolic blood pressure | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Systolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Diastolic blood pressure | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg
Heart rate | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in pulses/min.
Glucose concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood glucose levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Insulin concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood insulin concentration will be analyzed after an overnight fast by ELISA kit.
Blood glycated hemoglobin | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fasting blood glycated hemoglobin will be reported in percentage.
HOMA index | Clinical Investigation Day 1 and Clinical Investigation Day 2
  HOMA index will be calculated as follows: HOMA-IR = [fasting glucose (mmol/L) x fasting insulin (μU/ml)] / 22.5.
Total cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood total cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
HDL cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood HDL cholesterol levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL
LDL cholesterol | Clinical Investigation Day 1 and Clinical Investigation Day 2
  LDL cholesterol levels of participants in fasting condition will be analyzed by Friedewald formula and reported in mg/dL.
Triglyceride concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Triglyceride levels of participants in fasting condition will be analyzed by biochemical autoanalyzer and reported in mg/dL.
Hemogram concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Hemogram levels of participants in fasting condition will be analyzed by biochemical autoanalyzer.
Leptine | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood leptine concentration will be analyzed after an overnight fast by ELISA kit.
Adiponectin | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood adiponectin concentration will be analyzed after an overnight fast by ELISA kit.
MCP1 | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood MCP1 concentration will be analyzed after an overnight fast by ELISA kit.
Tumor necrosis factor alpha (TNF-alpha) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood TNF-alpha concentration will be analyzed after an overnight fast by ELISA kit.
C Reactive protein (CRP) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood CRP concentration will be analyzed after an overnight fast by ELISA kit.
Interleukin 10 (IL10) | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Blood IL10 concentration will be analyzed after an overnight fast by ELISA kit.
Albumin concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Albumin levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer.
Creatinine concentration | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Creatinine levels of participants in fasting condition will be analyzed in urine by biochemical autoanalyzer and reported in μmol/L.
Life quality | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Life quality of participants will be evaluated by SF-36 questionnaire.
chronotype | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Morningness-Eveningness Questionnaire (MEQ)
Level of hunger | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Hunger of participants will be analyzed by Hunger-Satiety Visual Analogue Scale (VAS). The minimum value of the scale is 0 mm and the maximum value is 100 mm. A reduction in hunger scale means better outcome.
Level of fullness | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Fullness of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in fullness scale means better outcome
Level of satisfaction | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Satisfaction sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. An incrementation in satisfaction scale means better outcome.
Want to eat something else | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Want to eat something else sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm. A reduction in want to eat something else scale means better outcome.
Thirst | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Thirst sensation of participants will be analyzed by Hunger-Satiety Visual Analogue Scale. The minimum value of the scale is 0 mm and the maximum value 100 mm.
Blood untargeted metabolomics | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Untargeted metabolomics will be analyzed in plasma and serum.
Urine untargeted metabolomics | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Untargeted metabolomics will be analyzed in urine.
Lipidomic | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Lipidomic will be analyzed in plasma and serum.
Depression | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Depression will be evaluated by Beck questionnaire.
Anxiety | Clinical Investigation Day 1 and Clinical Investigation Day 2
  Anxiety will be evaluated by Stai questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Idoia Ibero, PhD, Study Chair — Center for Nutrition Research; María Hernández, Study Chair — Center for Nutrition Research; Blanca Martínez, Study Chair — Center for Nutrition Research; Verónica Ciaurriz, Study Chair — Center for Nutrition Research; Carlos González, PhD, Study Chair — Center for Nutrition Research; Salomé Pérez, Study Chair — Center for Nutrition Research; Marta Cuervo, PhD, Study Chair — Center for Nutrition Research; Ana Lorente, Study Chair — Center for Nutrition Research; María Goñi, Study Chair — Center for Nutrition Research
Locations (1):
- Center for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No